CLINICAL TRIAL: NCT02300688
Title: An Open Label, Randomized, 2-sequence, 2-period, Single-dose Cross-over Study to Compare the Pharmacokinetics of Besifovir in Healthy Adult Volunteers
Brief Title: Bioequivalence Study to Compare the Pharmacokinetics of Besifovir in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ID_BVCL013
Record Dates: First submitted 2014-11-10; First posted 2014-11-25 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Period 1 (Treatment A) - Wash out - Period 2 (Treatment B)
  Interventions: Drug: Treatment A; Drug: Treatment B
- Arm 2 (Experimental): Period 1 (Treatment B) - Wash out - Period 2 (Treatment A)
  Interventions: Drug: Treatment A; Drug: Treatment B

INTERVENTIONS:
Drug: Treatment A — administration of 1 time administration of the test drug (Treatment A)
  Other Names: LB80380 maleate made by IDP
Drug: Treatment B — administration of 1 time administration of the reference drug (Treatment B)
  Other Names: LB80380 maleate made by LGLS

SUMMARY:
After administration of besifovir preparations different from each other to healthy subjects, the investigators evaluate equivalence of bioavailability of LB80331.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate equivalence of bioavailability of LB80331 preparations different. Following the randomly allocated sequence group administer the relevant test drug for 1 time according to the determined schedule of Treatment A and Treatment B in each of the periods.

ELIGIBILITY:
Inclusion Criteria:

1. Male whose age is 19 years or more and 55 years or less in full at the time of screening test
2. Subjects whose body mass index is 19 kg/m2 or more and 27 kg/m2 or less at the time of screening test
3. Subjects who listened to sufficient explanation of the purpose and contents of the Clinical Trial and characteristics of the test drug and spontaneously agreed to participate in the study in writing
4. Subjects who have ability and volition to participate in the Clinical Trial in the entire period of it

Exclusion Criteria:

1. Subjects who have clinically significant diseases or medical history of the diseases such as hepatobiliary, gastrointestinal, urinary, respiratory, cardiovascular system, musculoskeletal, endocrine system, neuropsychiatric disease, blood disease and tumor
2. Subjects who have hereditary problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
3. Subjects who have medical history of hypersensitivity to the drugs (aspirin, antibiotics) or have allergic diseases that require treatment
4. Subjects who were administered to investigational product within the past 60 days from the day of random allocation
5. Subjects who donated whole blood within the past 60 days from the day of random allocation or donated component blood within the past 30 days from the day of random allocation
6. Subjects who took the drug which needs doctor's prescription or oriental herbal medicine within the past 14 days from the day of random allocation or took over-the-counter drug within the past 7 days from the day of random allocation (Only, can be selected as subject according to decision of the investigator)
7. Subjects whose average drinking quantity per week exceeds alcohol 140g
8. Subjects whose average smoking quantity exceeds 20 cigarettes or subjects who cannot stop smoking during their hospitalization
9. Subjects whose average quantity of intake of grapefruit juice per day exceeds 4 glasses
10. Subjects whose systolic blood pressure is less than 90 mmHg or more than 140 mmHg or diastolic pressure is less than 60 mmHg or more than 100 mmHg at the time of screening test
11. Subjects whose AST, ALT, total bilirubin, γ-glutamyl transferasevalues in blood exceed 1.5 times of the upper limit of reference
12. Subjects whose Creatine phosphokinase value in blood exceeds 2.5 times of the upper limit of reference
13. Subjects whose glomerular filtration rate calculated from creatinine value in blood is less than 60 mL/min.
14. Subjects who do not show negative reaction in tests for hepatitis B, tests for hepatitis C, HIV test and tests for syphilis
15. Subjects who show positive reaction in urine drug screening test
16. Subjects who were decided to be not suitable for participation in the Clinical Trial by investigators for other reasons

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
AUClast | preodse, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15 hours post-dose
Cmax | preodse, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15 hours post-dose

SECONDARY OUTCOMES:
tmax | preodse, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15 hours post-dose
t1/2 | preodse, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15 hours post-dose
AUCinf | preodse, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 15 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Ryeol Kim, Ph D., Principal Investigator — Samsung Medical Center, Professor of department of clinical pharmacology